CLINICAL TRIAL: NCT00805961
Title: A Phase II Study of Concurrent Radiation Therapy, Temozolomide, and Bevacizumab Followed by Bevacizumab/Everolimus in the First-line of Treatment of Patients With Glioblastoma Multiforme
Brief Title: RT, Temozolomide, and Bevacizumab Followed by Bevacizumab/Everolimus in First-line Treatment of GBM
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SCRI Development Innovations, LLC (Other)
Collaborators: Genentech, Inc. (Industry); Novartis (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCRI CNS 10
Record Dates: First submitted 2008-12-09; First posted 2008-12-10 (Estimated); Results first posted 2012-09-21 (Estimated); Last update posted 2021-12-08 (Actual); Status verified 2021-11

CONDITIONS: Glioblastoma Multiforme
Keywords: Glioblastoma Multiforme; Radiation Therapy; Temozolomide; Bevacizumab; Everolimus
MeSH Terms: conditions — Glioblastoma | interventions — Radiotherapy; Combined Modality Therapy; Temozolomide; Bevacizumab; Everolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Intervention (Experimental): Combined Modality Treatment and Systemic Therapy
  Combined Modality Therapy - Radiation Therapy: 2 Gy/fraction, single daily fractions Monday-Friday, to total of 60 Gy Temozolomide: 75 mg/m2 by mouth daily Bevacizumab: 10 mg/kg IV every 2 weeks (Weeks 1, 3, 5, and 7)
  After the last dose of radiation, patients exhibiting an objective response, stable disease on MRI scan, or have stable/improved tumor-related symptoms will begin systemic therapy
  Systemic Therapy - Bevacizumab: 10 mg/kg IV every 2 weeks Everolimus: 10 mg by mouth daily
  Interventions: Radiation: Radiation therapy; Drug: Temozolomide; Drug: Bevacizumab; Drug: Everolimus

INTERVENTIONS:
Radiation: Radiation therapy — Radiation therapy, 2.0 Gy daily, 5 days per week by single daily dose, to a total of 60 Gy over 6 weeks
  Other Names: Combined Modality Treatment
Drug: Temozolomide — Temozolomide 75mg/m2 by mouth daily, beginning day 1 of radiation therapy and continuing through the last day of radiation therapy
  Other Names: Combined Modality Treatment
Drug: Bevacizumab — Bevacizumab 10mg/kg IV, every 2 weeks, beginning day 1 of radiation therapy
  Other Names: Combined Modality Treatment
Drug: Bevacizumab — Bevacizumab 10mg/kg IV, every 2 weeks, beginning Week 11
  Other Names: Systemic Therapy
Drug: Everolimus — Everolimus 10mg by mouth daily, beginning Week 11
  Other Names: Systemic Therapy

SUMMARY:
In this phase II trial the investigators plan to incorporate two targeted agents, bevacizumab and everolimus, into the first-line multimodality therapy of glioblastoma. In the first portion of the treatment, bevacizumab will be added to standard concurrent radiation therapy plus temozolomide. After completing radiation therapy, patients will continue treatment with the combination of bevacizumab and everolimus.

DETAILED DESCRIPTION:
Although this maintenance regimen departs from the standard treatment with single agent temozolomide, we feel this approach may add to the overall efficacy of treatment for the following reasons: 1) results with bevacizumab/everolimus in renal cell carcinoma suggest there is at least an additive efficacy when these drugs are used in combination; 2) the efficacy of single agent temozolomide following standard concurrent radiation therapy/temozolomide has not been proven, 3) the use of the three-drug maintenance program (i.e., bevacizumab/everolimus/temozolomide) would probably not be tolerated well on a chronic basis in this patient population; and 4) the bevacizumab/everolimus combination has potential advantages as a maintenance therapy, since it has been well tolerated for many months in patients with other malignancies.

ELIGIBILITY:
Inclusion Criteria:

* Age >=18 years.
* Histologically confirmed intracranial glioblastoma multiforme (WHO grade 4).
* Patients who have had partial or complete surgical debulking are eligible, as are those with inoperable glioblastoma.
* No previous treatment with radiotherapy or systemic therapy. Local therapy with a Gliadel wafer placed at the time of surgical debulking is permitted.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Adequate bone marrow function
* Adequate liver function:
* Serum creatinine <=1.5 x institutional ULN.
* Ability to swallow whole pills.
* Women of child-bearing potential must have a negative serum pregnancy test performed within 7 days prior to start of treatment. Women of child-bearing potential and men must agree to use adequate contraception (barrier method of birth control) while receiving study treatment and for 6 months after the last study treatment. Hormonal contraceptives are not acceptable as a sole method of contraception. Female patients must not breast feed.
* INR <1.3 or PT/PTT within normal limits in patients not receiving anticoagulation. However, patients receiving anticoagulation treatment with an agent such as warfarin or heparin are also eligible. For patients on warfarin, the INR should be measured prior to initiation of everolimus and monitored at least weekly, or as defined by the local standard of care, until INR is stable.
* Fasting serum cholesterol <=300 mg/dL OR <=7.75 mmol/L AND fasting triglycerides <= 2.5 x institutional ULN.

Exclusion Criteria:

* New York Heart Association (NYHA) grade II or greater congestive heart failure (see Appendix B) or symptomatic congestive heart failure.
* Inadequately controlled hypertension (defined as systolic blood pressure >150 mmHg and/or diastolic blood pressure >100 mmHg).
* History of myocardial infarction or unstable angina within 6 months prior to beginning study treatment.
* History of stroke or transient ischemic attack within 6 months prior to beginning study treatment.
* Significant vascular disease (e.g., aortic aneurysm, requiring surgical repair or recent peripheral arterial thrombosis) within 6 months prior to beginning study treatment.
* Prior history of hypertensive crisis or hypertensive encephalopathy.
* History of hemoptysis (>=1/2 teaspoon of bright red blood per episode) within 1 month prior to beginning study treatment.
* Evidence of bleeding diathesis or significant coagulopathy (in the absence of therapeutic anticoagulation).
* History of abdominal fistula or gastrointestinal perforation within 6 months prior to Day 1.
* Serious, non-healing wound, active ulcer, or untreated bone fracture.
* Proteinuria as demonstrated by urine dipstick for proteinuria >=2+. For patients with >=2+ proteinuria on dipstick urinalysis, a urine protein: creatinine (UPC) ratio will be determined or a 24-hour urine collection will be done. Patients with a UPC ratio <1 or a 24-hour urine protein <1 gram are eligible.
* Minor surgical procedures (excluding placement of a vascular access device), fine-needle aspirations, or core biopsies within 7 days prior to starting treatment.
* Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to starting protocol treatment or anticipation of need for major surgical procedure during the course of study treatment. Patients who have not recovered from the side effects of any major surgery are not eligible.
* Treatment with any investigational agents within 4 weeks of study entry.
* Chronic, systemic treatment with corticosteroids or other immunosuppressive agents. Topical or inhaled steroids are allowed.
* Other malignancies within the past 3 years except for adequately treated carcinoma in situ of the cervix or basal cell or superficial squamous (skin cell) carcinomas.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2009-01; Primary Completion 2009-10 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John D Hainsworth, M.D., Study Chair — SCRI Development Innovations, LLC
Locations (13):
- United States (13):
  - Clearview Cancer Institute, Huntsville, Alabama
  - Florida Cancer Specialists, Fort Myers, Florida
  - Northeast Georgia Medical Center, Gainesville, Georgia
  - Consultants in Blood Disorders and Cancer, Louisville, Kentucky
  - Center for Cancer and Blood Disorders, Bethesda, Maryland
  - Grand Rapids Clinical Oncology Program, Grand Rapids, Michigan
  - St. Louis Cancer Care, Chesterfield, Missouri
  - Research Medical Center, Kansas City, Missouri
  - Methodist Cancer Center, Omaha, Nebraska
  - South Carolina Oncology Associates, PA, Columbia, South Carolina
  - Tennessee Oncology, PLLC, Nashville, Tennessee
  - Peninsula Cancer Institute, Newport News, Virginia
  - Virginia Cancer Institute, Richmond, Virginia

REFERENCES:
- [Background] Hainsworth JD, Shih KC, Shepard GC, Tillinghast GW, Brinker BT, Spigel DR. Phase II study of concurrent radiation therapy, temozolomide, and bevacizumab followed by bevacizumab/everolimus as first-line treatment for patients with glioblastoma. Clin Adv Hematol Oncol. 2012 Apr;10(4):240-6. PMID 22706484

RESULTS

PARTICIPANT FLOW:
Groups:
- Overall Study: Radiotherapy administered in 2.0 Gy single daily fractions, Monday through Friday, to a total of at least 60 Gy. Temozolomide 75 mg/m2 orally daily and bevacizumab 10 mg/kg IV every 2 weeks, both beginning on day 1 of radiation therapy
Period: Modality Therapy
Arm/Group | Overall Study
Started | 68
Completed | 64
Not Completed | 4
Not completed — Withdrawal by Subject | 1
Not completed — Adverse Event | 1
Not completed — Disease Progression | 2
Period: Treatment-Free Interval
Arm/Group | Overall Study
Started | 64
Completed | 57
Not Completed | 7
Not completed — Adverse Event | 3
Not completed — Intercurrent Illness | 2
Not completed — Physician Decision | 1
Not completed — Lack of Efficacy | 1
Period: Maintenance Treatment
Arm/Group | Overall Study
Started | 57
Completed | 23
Not Completed | 34
Not completed — Lack of Efficacy | 13
Not completed — Intercurrent Illness | 7
Not completed — Adverse Event | 6
Not completed — Withdrawal by Subject | 5
Not completed — Symptomatic Deterioration | 2
Not completed — Withdrawn Consent | 1

BASELINE CHARACTERISTICS:
Arm/Group | Overall Study
Number analyzed (Participants) | 68
Age, Continuous [Median (Full Range); unit: years] | 59 [24 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29
  Male | 39
Region of Enrollment [Number; unit: participants]
  United States | 68

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS)
Description: Progression-free survival is defined as the duration of time from start of treatment to time of progression or death, whichever comes first.
Time Frame: 18 months
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Overall Study
Number analyzed (Participants) | 51
Months | 11.3 [9.3 to 13.1]

2. Secondary Outcome: Number of Participants Experiencing Toxicity After This Novel Multimodality Regimen
Description: The toxicity assessments were made according to the common terminology criteria for adverse events (CTCAE version 3.0) of the National Cancer Institute. Number of participants with Grade 1 to 5 adverse events are reported here.
Time Frame: 18 months
Measure: Count of Participants; unit: Participants
Arm/Group | Overall Study
Number analyzed (Participants) | 68
Participants | 53

3. Secondary Outcome: Overall Survival of Patients With Glioblastoma Multiforme Following Treatment With This Novel Multimodality Regimen
Description: Overall survival was defined as the interval from the first day of study treatment until the date of death.
Time Frame: 18 months
Measure: Number (95% Confidence Interval); unit: Months
Arm/Group | Overall Study
Number analyzed (Participants) | 68
Months | 13.9 [12.4 to NA] — At time of data analysis of 18 months, some patients were still alive making complete data collection to generate complete confidence interval.

4. Secondary Outcome: Objective Response Rate of Patients With Glioblastoma Multiforme Following Treatment With This Novel Multimodality Regimen
Description: Response to treatment was assessed by MRI using the MacDonald criteria based on the assessment of the MRI scan for measurable, evaluable, and new lesions. The objective response rate is defined as the proportion of patients with improvement and or decreased extent of lesions compared to baseline.
Time Frame: 18 months
Population: Only 51 patients had measurable tumor and were evaluable for response assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Overall Study
Number analyzed (Participants) | 51
Participants | 31

ADVERSE EVENTS:
Arm/Group | Overall Study
Serious Adverse Events (participants affected / at risk) | 32/68
Other Adverse Events (participants affected / at risk) | 53/68
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Overall Study (N=68)
Fatigue (General disorders) | 2 (2)
Myocardial Infarction (Cardiac disorders) | 1 (1)
Thrombotic Microangiopathy (Blood and lymphatic system disorders) | 1 (1) — Thrombotic Thrombocytopenic Purpura (TTP)
CNS Hemorrhage (Blood and lymphatic system disorders) | 1 (1)
Severe Epistaxis with Hematesis (Blood and lymphatic system disorders) | 1 (1)
Dehydration (Gastrointestinal disorders) | 1 (1)
Fever in absence of neutropenia (General disorders) | 1 (2)
Death (General disorders) | 2 (2)
Pain (General disorders) | 2 (3)
Cholecystitis (Hepatobiliary disorders) | 1 (1)
Pneumonia (Infections and infestations) | 3 (4)
Infection with Unknown ANC (Infections and infestations) | 1 (1)
Infection with Normal ANC (Infections and infestations) | 2 (2)
Febrile Neutropenia (Infections and infestations) | 1 (1)
Infection - Cellulitis (Infections and infestations) | 1 (1) — Herpes Orbital Cellulitis
Infection - Urinary Tract Infection (Infections and infestations) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1)
Necrotizing Fasciitis (Musculoskeletal and connective tissue disorders) | 1 (1)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 (1)
Seizure (Nervous system disorders) | 6 (7)
Cognitive Disturbance (Nervous system disorders) | 1 (1)
Neuropathy - Motor (Nervous system disorders) | 1 (1)
Somnolence (Nervous system disorders) | 1 (1)
CNS Ischemia (Nervous system disorders) | 2 (2)
Syncope (Nervous system disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Mental Status (Nervous system disorders) | 1 (1)
Confusion (Nervous system disorders) | 1 (1)
Neurology - Other (Nervous system disorders) | 1 (1) — Progressive Glioblastoma Multiforme
Renal Failure (Renal and urinary disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Pneumothorax (Surgical and medical procedures) | 1 (1)
Thrombosis/Thrombus/Embolism (Vascular disorders) | 10 (11)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Overall Study (N=68)
Neutropenia (Blood and lymphatic system disorders) | 4/57 (4) — Maintenance Treatment
Thrombocytopenia (Blood and lymphatic system disorders) | 11 (11) — Modality Treatment
Fatigue (General disorders) | 19 (19) — Modality Treatment
Hypertension (Cardiac disorders) | 4 (4) — Modality Treatment
Nausea/Vomiting (Gastrointestinal disorders) | 8 (8) — Modality Treatment
Stomatitis/Mucositis (Gastrointestinal disorders) | 7 (7) — Modality Treatment
Rash (Skin and subcutaneous tissue disorders) | 4 (4) — Modality Treatment
Thrombocytopenia (Blood and lymphatic system disorders) | 10/57 (10) — Maintenance Treatment
Fatigue (General disorders) | 27/57 (27) — Maintenance Treatment
Thrombosis/Embolism (Vascular disorders) | 8/57 (8) — Maintenance Treatment
Hypertension (Cardiac disorders) | 22/57 (22) — Maintenance Treatment
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 5/57 (5) — Maintenance Treatment
Proteinuria (Renal and urinary disorders) | 11/57 (11) — Maintenance Treatment
Stomatitis/Mucositis (Gastrointestinal disorders) | 7/57 (7) — Maintenance Treatment
Hyperlipidemia (General disorders) | 5/57 (5) — Maintenance Treatment
Diarrhea (Gastrointestinal disorders) | 4/57 (4) — Maintenance Treatment
Rash (Skin and subcutaneous tissue disorders) | 9/57 (9) — Maintenance Treatment
Nausea/Vomiting (Gastrointestinal disorders) | 3/57 (3) — Maintenance Treatment

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor can review/embargo results communications prior to public release for a period that is >60 days but ≤180 days from date submitted to sponsor, who may require changes to the communication in order to remove specifically identified confidential information (other than study data) and/or delay the proposed publication to enable the sponsor to seek patent protection for inventions. The PI may not publish its results until 18 mos. after the trial has been completed at all sites.